CLINICAL TRIAL: NCT03251079
Title: PRECISION Study: A Prospective, Multi-center Evaluation of Precision, Compression and Performance of a Novel Implanted Continuous Glucose Sensor Using a Next Generation Transmitter and Algorithm
Brief Title: PRECISION Study: Multi-center Study of Performance of a Novel Implanted CGM System Using a Next Generation Transmitter and Algorithm
Acronym: PRECISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0031
Record Dates: First submitted 2017-07-26; First posted 2017-08-16 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Continuous Glucose Monitoring Device (Experimental): Senseonics continuous glucose monitoring system
  Interventions: Device: Continuous glucose monitoring system

INTERVENTIONS:
Device: Continuous glucose monitoring system — Implanted continuous glucose monitoring system
  Other Names: Senseonics continuous glucose monitoring system

SUMMARY:
The purpose of this multi-center, prospective clinical study is to evaluate the performance of a novel, implanted Senseonics continuous glucose monitoring system (Senseonics CGM System) compared to Yellow Springs Instrument (YSI) glucose analyzer reference standard measurements using a next generation transmitter and algorithm. Other measures evaluated will be the effects of compression on performance and the safety of the Senseonics CGM system.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, age ≥18 years
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year
3. Subject has signed an informed consent form and is willing to comply with protocol requirements

Exclusion Criteria:

1. History of severe hypoglycemia in the previous 6 months. Severe hypoglycemia is defined as hypoglycemia resulting in loss of consciousness or seizure
2. History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months
3. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study.
4. A condition preventing or complicating the placement, operation, or removal of the Sensor or wearing of transmitter, including upper extremity deformities or skin condition.
5. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke in the past 6 months; uncontrolled hypertension (systolic>160 mm Hg or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign Premature Atrial Contractions (PACs) and Premature Ventricular Contractions (PVCs) allowed).

   Subjects with asymptomatic coronary artery disease (e,g, coronary artery bypass graft (CABG), stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from Cardiologist documented.
6. Hematocrit <30% or >55%
7. History of hepatitis B, hepatitis C, or HIV
8. Current treatment for a seizure disorder unless written clearance by neurologist to participate in study
9. History of adrenal insufficiency
10. Currently receiving (or likely to need during the study period):

    immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin); glucocorticoids (excluding ophthalmic or nasal). This exclusion does include the use of inhaled glucocorticoids and the use of topical glucocorticoids (over sensor site only); antibiotic for chronic infection (e.g. osteomyelitis, endocarditis)
11. A condition requiring or likely to require magnetic resonance imaging (MRI)
12. Known topical or local anesthetic allergy
13. Known allergy to glucocorticoids
14. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study. Conditions include but are not limited to psychiatric conditions, known current or recent alcohol abuse or drug abuse by subject history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
15. Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
16. The presence of any other active implanted device (as defined further in protocol)
17. The presence of any other CGM sensor or transmitter located in upper arm (other location is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (3):
- United States (3):
  - AMCR Institute Inc., Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitoring Device: Continuous glucose monitoring system: Implanted with Senseonics Eversense® Continuous Glucose Monitoring (CGM) System (Eversense® CGM System).
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring Device
Started | 36
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 32
  Black or African American | 1
  Asian | 2
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  More than One Race | 0
  Hispanic | 4
  Non-Hispanic | 31
Region of Enrollment [Number; unit: participants]
  United States | 35
Body Mass Index Class: Normal, Overweight, Obese [Mean (Standard Deviation); unit: kg/m2] | 28.2 (5.4)
Dominant Hand: Right, Left [Number; unit: participants]
  Right | 33
  Left | 2
Diabetes Type: Type I, Type II [Count of Participants; unit: Participants]
  Type I | 25
  Type II | 10
Years Since Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 26.0 (14.3)
Type of insulin therapy [Count of Participants; unit: Participants]
  None | 5
  Multiple daily injections | 11
  Continuous insulin infusion pump | 19
History of ketoacidosis and hypoglycemia in past 6 months [Count of Participants; unit: Participants]
  Ketoacidosis | 0
  Hypoglycemia | 0

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CGM System Through 90 Days Post-Insertion (MARD for Paired CGM and Reference Glucose Measurements)
Description: The effectiveness endpoint is the mean absolute relative difference (MARD), calculated for all paired Senseonics CGM System and reference glucose measurements through 90 days of Sensor use. MARD is defined as the average of absolute difference of paired Senseonics CGM System and reference glucose readings divided by the reference glucose reading (reference) for all reference glucose values, that is: MARD = ((SUM | (Glucose)sensor - (Glucose)reference | / (Glucose)reference ) / n ) x 100%, where n is the total number of CGM and reference glucose pairs after 90 days of sensor use (MARD is a percentage). Lower MARDs indicate higher (better) accuracy.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: Matched CGM and YSI pairs
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 35
Number analyzed (Matched CGM and YSI pairs) | 15170
percent | 9.6 [8.9 to 10.4]

2. Primary Outcome: Safety Endpoint
Description: Incidence of device-related or sensor insertion/removal procedure-related serious adverse events through 90 days post-insertion.
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: serious adverse events
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 35
serious adverse events | 0 [0.0 to 3.5]

ADVERSE EVENTS:
Time Frame: Through 90 days post Sensor insertion and sensor removal 10-day follow-up (up to 100 days)
Arm/Group | Continuous Glucose Monitoring Device
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Glucose Monitoring Device (N=35)
Other - Gastroenteritis (Gastrointestinal disorders) | 1
Hypoglycemic episode (Endocrine disorders) | 1
Other - Wound infection left foot, grade 4 (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring Device (N=35)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sensor Location Site - Pain/Discomfort (Skin and subcutaneous tissue disorders) | 2 (2)
Other - Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (5)
Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Pilonidal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Difficulty removing sensor (Skin and subcutaneous tissue disorders) | 1 (2)
Adhesive Patch Location Site - Irritation including redness, excoriation or ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Other - Darkening of skin at proximal end of sensor (Skin and subcutaneous tissue disorders) | 1 (2)
Other - Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Other - Dental Caries (General disorders) | 1 (1)
Other - Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT03251079/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03251079/SAP_001.pdf